CLINICAL TRIAL: NCT01627002
Title: A Phase 1, FIH, Double-blind, Randomised Placebo-controlled Study to Investigate the Safety, Tolerability, Immunogenicity and Pharmacokinetics of PA401, and the Effects of PA401 Following LPS Challenge, in Healthy Subjects
Brief Title: A Phase 1, First in Human Study to Investigate the Safety and Tolerability of PA401
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: ProtAffin Biotechnologie AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PA401/01; 2012-001189-14 (EudraCT Number)
Record Dates: First submitted 2012-06-12; First posted 2012-06-25 (Estimated); Results first posted 2013-09-23 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-07

CONDITIONS: Healthy Volunteers
Keywords: Phase 1; First in Human; Healthy Volunteers; Lipopolysaccharide Challenge

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PA401 (Experimental): PA401 is a potent inhibitor of neutrophil activation and transmigration under development as a novel parenteral anti-inflammatory therapy for respiratory indications such as chronic obstructive pulmonary disease (COPD) and Cystic Fibrosis (CF). PA401 is a genetically engineered and recombinantly expressed mutant of the bioactive form of human interleukin-8.
  Interventions: Biological: PA401
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: PA401 — Part A of Study: Subcutaneous, 0.1mg to 50mg, single ascending doses Part B of Study: Subcutaneous, up to 17.1mg, single dose
  Arms: PA401
Other: Placebo — Subcutaneous
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the safety, tolerability, immunogenicity and the way the body absorbs, distributes, breaks down and excretes various increasing single and multiple subcutaneous doses of PA401 in healthy subjects.

This study will also look at the effect of PA401 on inflammation in the lungs following an inhaled lipopolysaccharide (LPS) challenge (LPS is a bacterial cell wall fragment) and sputum induction (a procedure performed to help to cough up sputum (phlegm)) after a single subcutaneous dose of two dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged 18 to 65 years

Exclusion Criteria:

* Subjects with a clinically relevant medical history

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2012-05; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Ritter, MD, Principal Investigator — Quintiles, Inc.
Locations (1):
- Quintiles, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from June 2012 (first subject dosed) to April 2013 (last subject visit). The study was conducted in 2 parts; Part A was a single ascending dose study, Part B was a randomised placebo-controlled study to investigate the effect of a single dose of PA401 on sputum neutrophils following inhaled lipopolysaccharide challenge
Pre-assignment Details: In Part B, subjects were included at baseline if they had a baseline neutrophil level in induced sputum of ≤70%
Groups:
- Part B PA401 1.0 mg: PA401 1.0 mg was administered 30 minutes after lipopolysaccharide challenge
- Part B PA401 3.0 mg: PA401 3.0 mg was administered 30 minutes after lipopolysaccharide challenge
- Part B Placebo: Placebo was administered 30 minutes after lipopolysaccharide challenge
Period: Overall Study
Arm/Group | Part A PA401 0.1 mg | Part A PA401 0.3 mg | Part A PA401 1.0 mg | Part A PA401 3.0 mg | Part A PA401 10 mg | Part A Placebo | Part B PA401 1.0 mg | Part B PA401 3.0 mg | Part B Placebo
Started | 4 | 4 | 4 | 4 | 2 | 9 | 10 | 5 | 7
Completed | 4 | 4 | 4 | 4 | 2 | 9 | 10 | 5 | 7
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 27 | 22 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 22 | 49
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 27 | 22 | 49
Region of Enrollment [Number; unit: participants]
  United Kingdom | 27 | 22 | 49

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Adverse Events
Time Frame: up to 14 days post dose
Population: Safety analyses were performed on all subjects who receive a dose of PA401 or placebo and who had any post-dose measurements
Measure: Number; unit: Participants
Arm/Group | Part A PA401 0.1 mg | Part A PA401 0.3 mg | Part A PA401 1.0 mg | Part A PA401 3.0 mg | Part A PA401 10 mg | Part A Placebo | Part B PA401 1.0 mg | Part B PA401 3.0 mg | Part B Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 2 | 9 | 10 | 5 | 7
Participants | 3 | 3 | 4 | 2 | 2 | 3 | 7 | 5 | 4

2. Primary Outcome: Immunogenicity
Description: Anti-drug antibody data
Time Frame: Up to 28 days post dose
Population: Safety analyses were performed on all subjects who received a dose of PA401 or placebo and who had any post-dose assessments
Measure: Number; unit: participants
Arm/Group | Part A PA401 0.1 mg | Part A PA401 0.3 mg | Part A PA401 1.0 mg | Part A PA401 3.0 mg | Part A PA401 10 mg | Part A Placebo | Part B PA401 1.0 mg | Part B PA401 3.0 mg | Part B Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 2 | 9 | 10 | 5 | 7
participants
  Day 1 anti-drug antibody (ADA) positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 ADA positive and cross-reactive with IL-8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 1 Pre-existing IL-8 autoantibodies | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 15 ADA positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 15 ADA positive and cross-reactive with IL-8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 15 Pre-existing IL-8 autoantibodies | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 29 ADA positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 29 ADA positive and cross-reactive with IL-8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 29 Pre-existing IL-8 autoantibodies | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Pharmacokinetic Parameters: Maximum Observed Plasma Concentration (Cmax)
Time Frame: Up to 12 time-points up to 48 hours post dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A PA401 1.0 mg | Part A PA401 3.0 mg | Part B PA401 1.0 mg | Part B PA401 3.0 mg
Number analyzed (Participants) | 4 | 4 | 8 | 5
ng/mL | 1.88 (0.587) | 7.51 (2.64) | 1.29 (0.411) | 2.85 (0.805)

4. Secondary Outcome: Pharmacokinetic Parameters: Time of Occurrence of the Maximum Observed Plasma Concentration (Tmax)
Time Frame: Up to 12 time-points up to 48 hours post dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A PA401 1.0 mg | Part A PA401 3.0 mg | Part B PA401 1.0 mg | Part B PA401 3.0 mg
Number analyzed (Participants) | 4 | 4 | 8 | 5
hours | 2.75 (0.87) | 2.02 (0.40) | 2.09 (0.53) | 2.20 (1.10)

5. Secondary Outcome: Pharmacokinetic Parameters: Terminal Half-life (t1/2)
Time Frame: Up to 12 time-points up to 48 hours post dose
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A PA401 1.0 mg | Part A PA401 3.0 mg | Part B PA401 1.0 mg | Part B PA401 3.0 mg
Number analyzed (Participants) | 4 | 4 | 8 | 3
hours | 9.26 (2.57) | 8.44 (0.846) | 6.17 (1.79) | 10.1 (4.47)

6. Secondary Outcome: Pharmacokinetic Parameters: Area Under the Plasma Concentration-time Curve From Zero to Infinity
Time Frame: Up to 12 time-points up to 48 hours post dose
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Part A PA401 1.0 mg | Part A PA401 3.0 mg | Part B PA401 1.0 mg | Part B PA401 3.0 mg
Number analyzed (Participants) | 3 | 4 | 7 | 3
ng.h/mL | 23.9 (9.72) | 93.2 (12.1) | 12.2 (3.82) | 29.3 (5.66)

7. Primary Outcome: Assessment of the Effect of PA401 on Induced Sputum Total Neutrophils
Description: Induced sputum was collected 6 hours after lipopolysaccharide challenge (5.5 hours following dosing) and assessed for neutrophils
Time Frame: 5.5 hours post dose
Measure: Least Squares Mean (95% Confidence Interval); unit: x10e6 cells/g
Arm/Group | Part B 3.0 mg PA401 | Part B 1.0 mg PA401 | Part B Placebo
Number analyzed (Participants) | 5 | 10 | 7
x10e6 cells/g | 11.6882 [2.8474 to 20.5290] | 7.7274 [1.4038 to 14.0511] | 12.7241 [5.1749 to 20.2733]

8. Secondary Outcome: Assessment of the Effect of PA401 on Induced Sputum Percentage Neutrophils
Description: as for outcome 7
Time Frame: 5.5 hours post dose
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of total cells
Arm/Group | Part B 3.0 mg PA401 | Part B 1.0 mg PA401 | Part B Placebo
Number analyzed (Participants) | 5 | 10 | 7
percentage of total cells | 32.9429 [26.0955 to 39.7902] | 36.7007 [31.7343 to 41.6670] | 34.3856 [28.4360 to 40.3352]

ADVERSE EVENTS:
Time Frame: Up to 14 days post dose
Description: Adverse events were monitored by the clinical staff asking non-leading questions during the period of confinement to the clinic.
Arm/Group | Part A PA401 0.1 mg | Part A PA401 0.3 mg | Part A PA401 1.0 mg | Part A PA401 3.0 mg | Part A PA401 10 mg | Part A Placebo | Part B PA401 1.0 mg | Part B PA401 3.0 mg | Part B Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 1/2 | 0/9 | 0/10 | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 3/4 | 3/4 | 4/4 | 2/4 | 2/2 | 3/9 | 7/10 | 5/5 | 4/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A PA401 0.1 mg (N=4) | Part A PA401 0.3 mg (N=4) | Part A PA401 1.0 mg (N=4) | Part A PA401 3.0 mg (N=4) | Part A PA401 10 mg (N=2) | Part A Placebo (N=9) | Part B PA401 1.0 mg (N=10) | Part B PA401 3.0 mg (N=5) | Part B Placebo (N=7)
Atrial Fibrillation (Cardiac disorders) | 0/3 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A PA401 0.1 mg (N=4) | Part A PA401 0.3 mg (N=4) | Part A PA401 1.0 mg (N=4) | Part A PA401 3.0 mg (N=4) | Part A PA401 10 mg (N=2) | Part A Placebo (N=9) | Part B PA401 1.0 mg (N=10) | Part B PA401 3.0 mg (N=5) | Part B Placebo (N=7)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (12) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection Site Erythema (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 2 (2)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection Site Reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-Reactive Protein Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Disturbance In Attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
Part B of the study was terminated early which led to a small number of subjects analyzed. Pharmacokinetic parameters were not calculated for Part A 0.3mg and 10 mg PA401

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After completion of the study, the Investigator may prepare a joint publication with the Sponsor. The Investigator must undertake not to submit any part of the individual data from this protocol for publication without prior consent of the Sponsor at a mutually agreed time.